CLINICAL TRIAL: NCT01146067
Title: Bioequivalence Study of Rivastigmine 1.5 mg Capsules (Test)of Dr.Reddy's Laboratories Limited Versus Exelon (Reference),Administered as 1 x 1.5 mg Capsule Under Fasting Conditions
Brief Title: Bioequivalence Study of Rivastigmine 1.5 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sr.Manager -R&D, Dr.Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30496
Record Dates: First submitted 2010-02-10; First posted 2010-06-17 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivastigmine (Experimental): Rivastigmine capsules 1.5 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Rivastigmine
- Exelon (Active Comparator): Exelon 1.5 mg capsules of Novartis
  Interventions: Drug: Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine — Rivastigmine capsules 1.5 mg
  Other Names: Exelon 1.5 mg capsules

SUMMARY:
This is a bioequivalence study of Rivastigmine 1.5 mg capsules and Exelon Administered as 1.5 mg capsule in Healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
Single center, bioequivalence, open-label, randomized, 2-way crossover study administered as 1 x 1.5 mg capsule in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study will be members of the community at large.
* The recruitment advertisements may use various media types (e.g. radio, newspaper, Anapharm Web site, Anapharm volunteers' database). Subjects must meet all of the following criteria in order to be included in the study:

  * Male or female, smoker or non-smoker, 18 years of age and older.
  * Capable of consent.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis H, hepatitis C, or HN at screening.
* BCG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* BMI2: 30.0.
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (l Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to rivastigmine or other related drugs.
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine)within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological,endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption or hormonal contraceptives.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food energy, intolerance, restriction or special diet that could, in the opinion of the Medical Sub-Investigator, contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptive) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 300 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* History of ulcer disease.
* History of asthma or obstructive pulmonary disease.
* Use of any nonsteroidal anti-inflammatory drugs (e.g. Motrin®, Advil®, within 14 days prior to drug administration.
* History of seizures, urinary obstruction or benign prostatic hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D, Principal Investigator — Anapharm Inc, Canada